CLINICAL TRIAL: NCT06774014
Title: Heart Failure in Patients With Diabetes: Cells, Crosstalk and Consequences
Status: Recruiting | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Klaus K Witte, MD, Senior Lecturer in Cardiology, University of Leeds
Other Study IDs: 2024-NCT37; RE_23_130040-3 (Other Grant/Funding Number: British Heart Foundation); CD25/177037 (Other: LTHT)
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus Type 2; Heart Failure; HFrEF - Heart Failure With Reduced Ejection Fraction; HFpEF - Heart Failure With Preserved Ejection Fraction
Keywords: Crosstalk; Metabolomics; Proteomics; Fat; Skeletal muscle; Vascular function; Autonomic function; Endothelial function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood, fat, muscle, endothelial cells
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- HFrEF-DM: People with heart failure due to reduced ejection fraction without diabetes mellitus
- HFrEF+DM: People with heart failure due to reduced ejection fraction who also have diabetes mellitus
- HFpEF-DM: People with heart failure with preserved ejection fraction without diabetes mellitus
- HFpEF+DM: People with heart failure with preserved ejection fraction who also have diabetes mellitus
- DM: People who have diabetes mellitus but do not have heart failure
- Control: People who have neither heart failure nor diabetes mellitus

SUMMARY:
This will be an observational study to explore differences in pathophysiology between groups of people with and without heart failure (HF) (reduced and preserved ejection fraction) and with and without diabetes mellitus (DM) with a particular focus on cross-talk (fat, muscle, vascular tissue and the heart). The investigators will invite 600 people to partcipate (100 with HFrEF+DM, 100 with HFpEF+DM, 100 with HFpEF-DM, 100 with HFrEF-DM, 100 with DM, 100 without either HR or DM). Special heart scans, exercise testing, blood testing, testing of the automatic nervous system will be performed and in some, samples of fat and muscle and endothelial cells will be collected.

These data will be used to create a cohort of well phenotyped patients with a variety of comprehensively collected clinical information, a cell atlas, and a comprehensive assessment of metabolomics, proeomics and cross-talk in between tissues, allowing comparisons between each group.

DETAILED DESCRIPTION:
Heart failure is a leading cause of mortality and morbidity worldwide, and is characterized by symptoms such as shortness of breath, peripheral oedema and impaired exercise capacity due to structural or functional heart disease. The condition is associated with impaired longevity, high levels of morbidity (poor quality of life) and enormous costs for the healthcare system. In the western world, approximately 1-2% of the population suffer from heart failure, increasing to over 10% of people over the age of 70. The prognosis of patients with severe heart failure is similar to that of patients with cancer.

Diabetes mellitus is reaching pandemic proportions across the globe. A condition previously characterised simply as a relative or absolute deficiency of insulin and diagnosed by elevated sugar levels in the bloodstream, it is now much better understood as a syndrome of impaired glucose tolerance accompanied by a range of metabolic abnormalities that can be observed in all tissues of the body. This metabolic remodelling is accompanied by higher risks of chronic disease particularly cardiovascular disease including atherosclerosis but also, even in the absence of coronary artery disease, a considerable increase in the risk of heart failure.

These two morbid and life-limiting illnesses commonly occur together, each worsening the other in a synergistic relationship that leads to greater symptoms, resistance to therapies and shorter longevity.

Further detail on how these diseases interact is urgently required. However, in addition to understanding the clinical impacts on patients, in order to focus existing therapies and develop new options, it is necessary to understand how these diabetes mellitus an heart failure interact at a metabolic level, which cellular-based pathways are affected and how these lead to abnormal cellular function, and thereby to tissue and organ dysfunction. Further understanding of how communication between tissues contributes to the overall pathophysiology is required.

The present investigation will therefore be a single-centre non-randomised, observational study involving an unselected but highly phenotyped cohort of patients with and without heart failure and with and without type 2 diabetes mellitus and controls without disease. Patients will be recruited from heart failure and diabetes clinics and controls will be identified from these patients' carers and their relatives through direct contact and advertisements in outpatient departments.

Participants will undergo cardiac ultrasound, exercise testing, assessments of lung function, non-invasive haemodynamics, autonomic function, hand and leg muscle strength, and lung function assessment along with blood testing, longer term glucose monitoring and blood sampling. A small sample of fat and muscle will be collected. A subgroup will undergo an MRI scan of the heart and their thigh muscles. Participants' involvement will end at that point although they will continue to be monitored using their digital records on an annual basis for up to 10 years to gain information on the prognostic value of the metabolic and haemodynamic testing.

Tissue and blood samples will be coded and stored in a Human Tissue Authority-approved freezer until analysis following which they will be related to clinical variables with the aim of identifying mechanisms by which metabolic disease (in this case diabetes mellitus) influences the progression of heart failure with the long term objective of informing the development of more effective treatment strategies.

The present investigation will allow the investigators to advance the understanding of how metabolic disease and heart failure interact with the goal of developing targeted interventions that could open new treatment avenues.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Ability to provide written informed consent
* Persons who are legally competent and mentally able to follow the instructions of the study staff

Exclusion Criteria:

* Anaemia Hb <8 mg/dl
* Patients with acute infectious diseases (e.g. pneumonia)
* Patients with heart failure due to sepsis
* People with acute myocardial ischemia, which is manifested, for example, by angina pectoris or ECG changes under stress
* Patients with acute liver or kidney failure or severe COPD (FEV1<1.0)
* Pregnant and breastfeeding women
* People who are institutionalized on official or court orders
* People who are dependent or employed by the sponsor or investigator
* Taking study medication (of an investigational drug) 30 days before the start of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People attending heart failure clinics, diabetes clinics (either secondary or primary care) or control subjects attending hospital with relatives or accumulated from the community by word of mouth or advertisement.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Study primary endpoint | 5 years
  Are there differences in skeletal muscle cellular metabolism assessed by mass spectrometry-based metabolomics and lipidomics between the two phenotypes of heart failure compared with controls and what influence does diabetes mellitus have?

SECONDARY OUTCOMES:
Secondary outcome 1 | 5 years
  How does T2DM influence intercellular communication to promote the progression of HF
Secondary outcome 2 | 5 years
  Are there correlations between abnormalities in these cells and cardiac abnormalities, patient symptoms and clinical outcomes?
Secondary outcome 3 | 5 years
  What metabolic pathways are abnormal in people with heart failure, diabetes mellitus and both?
Secondary outcome 4 | 5 years
  Can we identify using metabolomics, a substrate or compound that underlies the metabolic abnormalities?
Secondary outcome 5 | 5 years
  Does organ 'cross-talk' have a negative influence on the functions of skeletal muscle, fat, platelets and clotting function, and cardiac function?
Secondary outcome 6 | 5 years
  Is autonomic activation reflected in metabolic abnormalities in HFrEF or HFpEF?
Secondary outcome 7 | 5 years
  Is lung function, especially that of the diaphragm and smooth muscle of the medium-sized bronchioles reflective of the metabolic abnormalities and how do these relate to the two major HF phenotypes?
Secondary outcome 8 | 5 years
  Do the laboratory data describing muscle and fat metabolomics relate to clinical variables and prognosis?
Secondary outcome 9 | 5 years
  Is cardiac contractility impairment as measured by cardiac magnetic resonance related to the tissue-based metabolic abnormalities and can we identify different subgroups of contractile function within the heart failure and diabetes groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
An anonymised version of the database and the samples will be available to other researchers including outside of the University of Leeds in response to a reasonable request and confirmation of appropriate data protection policies and a mutual data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after the end of the study
Access Criteria: Requests to be made to the Trial Management Group

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT06774014/Prot_SAP_000.pdf